CLINICAL TRIAL: NCT06225817
Title: The Impact of Open-label Placebo on Sleep and Pain Modulation
Brief Title: Placebo Impacts Sleep and Pain Modulation in Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HP-00105618
Record Dates: First submitted 2024-01-16; First posted 2024-01-26 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain; Headache
MeSH Terms: conditions — Chronic Pain; Headache

STUDY DESIGN:
Intervention Model Description: This is a longitudinal parallel randomized clinical trial with chronic headache participants randomly assigned to either 1) OLP+Expectations management; 2) OLP alone; or 3) Standard of care. To examine how baseline chronic pain and sleep patterns could have impacted the effects of OLP, we will deep-phenotype participants based on their sleep profiles and fluctuations in their chronic pain characteristics via a 2-day phenotyping phase. Following the 2-day phenotyping phase, participants will enter a 45-day intervention phase. The nature of the participation will be voluntary. Namely, participants can withdraw during trial from the study without any consequences.
Who Masked: Outcomes Assessor
Masking Description: There is no masking in the study. Both the participants and the experimenter know that the participants will be taking open-label placebos.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Open label placebo only arm (Experimental): Participants who are assigned to the OLP group will be given a bottle of OLP pills. They will be asked to take one pill per day for 45 days. They will be introduced to placebo effects and the therapeutic potential of using open-label placebo for chronic pain management and sleep improvement.
  Interventions: Dietary Supplement: Open-label placebo pills
- Wait-list arm (No Intervention): Participants in the wait-list group will not receive OLP pills until the end of the 45-day monitoring period. Therefore, the 45 days without OLP will serve as an no intervention comparators relative to the OLP group.
- Open label placebo + expectation management (Experimental): Participants assigned to this arm will complete an 1 hour discussion about their expectations towards open-label placebo intervention. After that, they will continue with the 2-day run-in period and 45-day intervention. They will be asked to take 1 open-label placebo pill per day, for a total of 45 days.
  Interventions: Dietary Supplement: Open-label placebo pills

INTERVENTIONS:
Dietary Supplement: Open-label placebo pills — The placebo pills in this study are empty capsules without any ingredients inside. The capsules are made of microcrystalline cellulose.
  Other Names: Zeebo pills
  Arms: Open label placebo + expectation management; Open label placebo only arm

SUMMARY:
The goal of this free-choice parallel design clinical trial is to examine the potential beneficial effects of using open-label placebo (OLP) in improving chronic pain related outcomes and sleep quality in people with temporomandibular disorders. This study will enroll a cohort of participants with temporomandibular disorders (TMD) which lasts for more than 3 months. The main questions it aims to answer are:

1. Will participants with TMD be more likely to take open-label placebo pills if they are introduced to the effects of placebo (e.g., going through an expectation management session)?
2. Will taking open-label placebo plus expectation management improve chronic pain related outcomes, such as chronic pain intensity, interference, levels of anxiety and depression, in the cohort of TMD?
3. Will open-label placebo plus expectation management improve sleep quality in participants suffering from TMD?

To answer the above questions, participants with TMD will be randomly assigned to three groups: 1. Open-label placebo plus expectation management group, where participants will complete a 1-hour discussion session about their expectations toward open-lable placebo intervention, and then take 1 open-labe placebo pill per day for a total of 45 days. 2. Open-label placebo only group where participants will be asked to take open-label placebo pills, one pill per day, for a total of 45 days. 3. standard of care group where participants will maintain their usual care without introducing open-label placebo to them during the 45 days monitoring. Researchers will compare the chronic pain intensity, interference, mood, anxiety, and sleep quality between the open-label placebo group and the wait-list group. Daily chronic pain will be measured using visual analog scale (VAS) ranging from 0=no pain at all to 100=maximum tolerable pain. Chronic pain interference using Patient-Reported Outcomes Measurement Information System (PROMIS) pain interference and pain behavior. Anxiety and depression will be measured using PROMIS-anxiety, and PROMIS-depression scales respectively. Finally, sleep quality will be quantified using the objective measurement Motion Watch during the 45 days intervention and monitoring. In order to have a rigorous measurement of the baseline pain and sleep fluctuation, this study will include a 7-day phenotyping period before the starting of the 45-day intervention and monitoring. During the 7-day phenotyping period, participants will record their daily chronic pain and sleep quality using polysomnography.

DETAILED DESCRIPTION:
This is a longitudinal parallel randomized clinical trial with TMD participants randomly assigned to either 1) the open-label placebo (OLP) + expectations management group, 2) OLP only, and 3) the standard of care group. To examine how baseline chronic pain and sleep patterns could have impacted the effects of OLP, we will deep-phenotype participants based on their sleep profiles and fluctuations in their chronic pain characteristics via a 2-day phenotyping phase. Following the 2-day phenotyping phase, participants will enter a 45-day intervention phase. The nature of the participation will be voluntary. Namely, participants can withdraw during trial from the study without any consequences.

Phenotyping phase (2-day) The phenotyping phase includes an in-person visit and a 2-day at-home monitoring period. During the in-person visit, after signing the informed consent form with the trained staff, participants will complete a heat pain sensitivity test using a 30mmx30mm Advanced Thermal Stimulator (ATS) via the Medoc Pathway system (Medoc Advanced Medical Systems, Medoc Ltd., Israel). Painful and non-painful stimuli will be delivered to the ventral forearm of the non-dominant hand.

After the in-person visit, participants will enter a 2-day daily monitoring period, where their daily pain expectations, pain experience fluctuations, and sleep diaries will be assessed in real time and in their natural environment using the Ecological Momentary Assessment (EMA) method. Sleep profiles will be assessed using polysomnography to obtain natural sleep architectures, including the duration of different sleep stages, sleep efficiency, breathing, and body movement during sleep.

Free-choice OLP intervention Immediately following the phenotyping phase, participants will return to the laboratory before entering the 45-day intervention phase. Participants will be randomized to either 1. OLP+expectations management, 2. OLP alone, and 3. Standard of care groups. Participants in the two OLP groups will receive a bottle of 45 OLP pills. According to the free-choice paradigm, participants in the OLP group are allowed to choose whether to take the pills each day during the intervention. This paradigm maximizes participant benefit because it provides the option of "not" taking the placebo pills. Participants in the wait-list group will not receive OLP pills until the end of the 45-day monitoring period.

ELIGIBILITY:
Inclusion Criteria:

* Age ( 18-88 years old)
* English speaker (written and spoken)
* TMD for at least 3 months
* Grade Chronic Pain Scale (GCPS) ≥1
* Smartphone/text messaging capability

Exclusion Criteria:

* Present or past degenerative neuromuscular disease
* Cardiovascular, neurological diseases, pulmonary abnormalities, kidney disease, liver disease, history of cancer within past 3 years
* Any personal (or family first degree) history of mania, schizophrenia, or other psychoses
* Severe psychiatric condition (e.g. schizophrenia, bipolar disorders, autism) leading to hospitalization within the last 3 years.
* Lifetime alcohol/drug dependence or alcohol/drug abuse in past 3 months
* Pregnancy or breast feeding
* Impaired or uncorrected hearing

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Chronic pain intensity | Daily over the 45 days
  Chronic pain intensity will be measured using visual analog scale ranging from 0=no pain at all to 100=maximum tolerable pain
Sleep efficiency | Daily over the 45 days
  Sleep efficiency will be measured using actigraphy motion watch ranging from 0%=efficient at all to 100% maximum efficient sleep

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Baltimore School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data including the daily monitoring of chronic pain and sleep quality will be shared after the publication of the study results.
Supporting Information: Study Protocol, SAP, ICF